CLINICAL TRIAL: NCT02570516
Title: Comparison of Colonoscopy With Virtual Chromoendoscopy Using 3rd Generation NBI System to Chromoendoscopy With Indigo Carmine in Lynch Patients.
Brief Title: NBI Versus Indigo Carmine During Colonoscopy in Lynch Syndrome
Acronym: LYNCH-CHROMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: ARC Foundation for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: P140108; 2015-A00552-47 (Other Grant/Funding Number: ANSM)
Record Dates: First submitted 2015-09-30; First posted 2015-10-07 (Estimated); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Lynch Syndrome
Keywords: Indigo carmine chromoendoscopy; Narrow band imaging; Colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Indigo carmine colonoscopy (Active Comparator): Colonoscopy using indigo carmine is performed in second place
  Interventions: Procedure: Colonoscopy
- NBI colonoscopy (Experimental): Colonoscopy using NBI is performed in first place
  Interventions: Procedure: Colonoscopy

INTERVENTIONS:
Procedure: Colonoscopy — A double colonoscopy is performed in a back-to-back design using NBI chromoendoscopy then indigo carmine in each patient.

SUMMARY:
This study compares two colonoscopy techniques (with Narrow Band Imaging versus with indigo carmine chromoendoscopy) in patients having Lynch Syndrome

DETAILED DESCRIPTION:
Chromoendoscopy using indigo carmine dye is recommended every 1 to 2 years in patients having Lynch Syndrome (LS). However, it is a time-consuming procedure, requiring a prior learning and has an additional cost, the reason why it is not yet systematically practiced in all endoscopy centers. The "Narrow Band Imaging" (NBI) is a recent virtual chromoendoscopy technique using optical filters at the light source of the endoscope to highlight the vascular structures of the mucosa by pressing a button. NBI is currently used to better characterize dysplasia lesions in the esophageal, gastric, and colon mucosa. A new generation (3rd generation) of NBI is currently available on some endoscopes, it can deliver more brightness and contrast, and could allow for better detection of flat lesions. Until today, no study has directly compared colonic chromoendoscopy with Indigo carmine to virtual chromoendoscopy with NBI (3rd generation) in LS patients. The hypothesis that this research aims to verify is that the new generation NBI system might do at least as well as indigo carmine in colonic adenoma detection in LS. This study aims to compare colonoscopy with virtual chromoendoscopy using 3rd generation NBI system to chromoendoscopy with indigo carmine in LS patients, in a back-to-back, prospective non inferiority design, in which all patients will have both techniques in the following order: NBI first followed by Indigo carmine.

ELIGIBILITY:
Inclusion Criteria:

* Lynch Syndrome with an identified mutation in one of the genes MutL Homolog 1 (MLH1), MutL Homolog 2 (MLH2), MutS homolog6 (MSH6), PMS2 or epithelial cellular adhesion molecule (EpCAM)
* Age between 18 and 80
* Indication of a screening colonoscopy

Exclusion Criteria:

* Any sign of intestinal occlusion contra-indicating bowel preparation
* History of total or subtotal colectomy
* Any serious medical condition contra-indicating colonoscopy under general anesthesia
* Pregnant or breast feeding women
* Any coagulation disorder contra-indicating biopsies or endoscopic resections
* Any history of hypersensitivity to indigo carmine
* Adults subject to a legal protection measure (guardianship or curatorship)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Number of adenomas and / or adenocarcinoma detected during each procedure (NBI vs Indigo carmine) | procedure time
  The adenoma detection rate (number of adenoma and/or adenocarcinoma) of NBI and the additional adenoma detection rate of indigo carmine.

SECONDARY OUTCOMES:
All neoplastic lesions detected during colonoscopy | procedure time
  Collect the number, size, location, endoscopic (Paris Classification) and anatomo-pathologic aspect (adenoma, hyperplastic polyp, adenocarcinoma) of all detected lesions with their respective prevalence.
Cost of each procedure (NBI vs Indigo carmine) | Procedure time
  Evaluate the cost of each procedure including therapy.
Duration of each procedure (NBI vs Indigo carmine) | Procedure time
  Evaluate the duration of each procedure (with and without endoscopic therapy).
Number of subject with adverse events as mesure of safety. | One month after colonoscopy
  Followed a month post colonoscopy to evaluate the occurrence of undesirable events

CONTACTS AND LOCATIONS:
Overall Officials: CHRISTOPHE CELLIER, MD, PHD, Principal Investigator — Hopital europeen Georges Pompidou
Locations (7):
- France (7):
  - HCL - Hôpital Edouard-Herriot, Lyon, Auvergne-Rhône-Alpes
  - CHRU de Tours - Hôpital Trousseau, Chambray-lès-Tours, Centre-Val de Loire
  - CHU Nantes - Hôtel-Dieu, Nantes, Pays de la Loire Region
  - AP-HP - Hôpital Européen Georges-Pompidou, Paris
  - AP-HP - Hôpital Saint-Antoine, Paris, Île-de-France Region
  - AP-HP - Hôpital Cochin, Paris, Île-de-France Region
  - Institut Gustave-Roussy, Villejuif, Île-de-France Region

REFERENCES:
- [Derived] Cellier C, Perrod G, Colas C, Dhooge M, Saurin JC, Lecomte T, Coron E, Rahmi G, Savale C, Chaussade S, Bellanger J, Dray X, Benech N, Le Rhun M, Barbieux JP, Pereira H, Chatellier G, Samaha E. Back-to-Back Comparison of Colonoscopy With Virtual Chromoendoscopy Using a Third-Generation Narrow-Band Imaging System to Chromoendoscopy With Indigo Carmine in Patients With Lynch Syndrome. Am J Gastroenterol. 2019 Oct;114(10):1665-1670. doi: 10.14309/ajg.0000000000000386. PMID 31498154